CLINICAL TRIAL: NCT01434758
Title: Evaluating Diagnostics for Paediatric Tuberculosis by Blood Culture
Status: Completed | Type: Observational
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: National Children's Hospital, Vietnam (Other)
Responsible Party: Sponsor
Other Study IDs: 09TB
Record Dates: First submitted 2011-04-06; First posted 2011-09-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Tuberculosis Infection
Keywords: Mycobacterium tuberculosis; Culture yield
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * sputum
  * gastric aspirate
  * blood
  * urine
  * cerebrospinal fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children: Children age 0-15 years presenting to NHP thought to have TB infection

SUMMARY:
Detection of M. tuberculosis in clinical specimens of children has a low sensitivity because specimens are either difficult to collect or contain low levels of M. tuberculosis. Diagnostic criteria are non-specific and culture confirmation is challenging, as sputum samples are not often obtainable from small children and specimens typically have low yield. Although children are typically thought to have paucibacillary disease, they are at greater risk for dissemination of TB. This may allow for detection of Mycobacterium tuberculosis from other bodily fluids than sputum or gastric aspirate, including blood and urine. Unfortunately, little is known about the overall yield from these various specimens. From pilot data collected among adults and children in Tugela Ferry, we know that it is feasible to collect and test various bodily fluid specimens for TB culture. This study aim to test the hypothesis that blood and urine cultures will detect Mycobacterium tuberculosis from children suspected of disseminated TB, and that a proportion of these non-sputum bodily fluids will detect both drug-susceptible and drug-resistant tuberculosis when sputum or gastric culture does not.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major cause of morbidity and mortality among children in developing nations. Symptom-based diagnostic criteria are non-specific and culture confirmation is challenging, as sputum samples are often believed to be to too cumbersome to obtain from small children and specimens typically have low yield due to the paucibacillary nature of pediatric TB. Culture confirmation may be obtained in as few as 10% of cases of suspected pediatric TB. For these reasons, the true extent of the (drug-resistant) TB epidemic in children is unknown. Thus, either clinicians begin empiric treatment without diagnosis or no treatment is given at all. Current laboratory methods, if available at all in resource poor settings, employ smears from expectorated sputa or gastric aspirates which have low sensitivity in children. While more rapid diagnostic techniques such as PCR based tests have been developed, there is still poor sensitivity in children. Improving the diagnosis of pediatric TB must focus on better efforts, including more aggressive strategies to uncover disseminated disease.

Culture confirmation of disseminated disease can be obtained from blood, urine, cerebrospinal fluid (CSF), peritoneal and pleural fluid, or purulent material from lymph node aspirates, abscesses or otorrhea. Unfortunately, little is known about the overall yield from these various specimens in children. From pilot data collected among children at NHP, we know that it is feasible to collect and test various bodily fluid specimens for TB culture.

Although WHO guidelines encourage body fluid collection in order to make a diagnosis of TB in children, at present in NHP, blood and urine cultures are not obtained for mycobacterial culture. However, this study seeks to demonstrate that routine investigation of blood and urine will augment the yield of traditional sputum culture for children in whom disseminated disease is more likely. Improved culture confirmation will allow DST and a more accurate description of the drug-resistant TB epidemic for children in the region.

ELIGIBILITY:
Inclusion Criteria:

* Aged 0-15, presenting at NHP;
* Unexplained fever for more than 2 weeks; and
* Any form of TB suspected based on at least two of the following findings:

  * unexplained cough for more than 2 weeks
  * radiographic findings suggestive of tuberculosis.
  * failure to thrive/weight loss
  * enlarged non-tender lymph nodes or lymph node abscess, especially of the neck
  * signs of meningitis with prodromal stage of at least one week
  * HIV positive
  * malnourished
  * TB contact history
  * Clinical judgment treating doctor.
* Relevant material (sputum or gastric aspirate, blood, and urine) available for microbiological diagnosis.
* Informed consent obtained from the patient's legal guardian(s).

Exclusion Criteria:

* Age >15 years
* Diagnosed or treated for TB in the past year, received drugs effective against TB in last 3 months.
* Clinical contra-indications to collect the required study specimens

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population is children aged 0-15 years presenting to NHP thought to have TB infection according to inclusion criteria listed in this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of TB culture | At baseline - day 1 of study
  Number of positive TB cultures versus number of positive TB direct smears for expectorate and/or gastric aspirate.
Diagnostic yield of TB culture | At baseline - day 1 of study
  Number of positive TB cultures versus number of positive MODS cultures for expectorate and/or gastric aspirate.
Diagnostic yield of urine versus expectorate or gastric aspirate for TB culture | At baseline - day 1 of study
  Number of positive TB cultures in urine versus expectorate and/or gastric aspirate.

CONTACTS AND LOCATIONS:
Overall Officials: Heiman F Wertheim, PhD, Principal Investigator — Oxford University Clinical Research Unit - Hanoi
Locations (1):
- National Hospital of Pediatrics, Hanoi, Hanoi, Vietnam

REFERENCES:
- See also: OUCRU studies public site — http://www.oucru.org/index.php?option=com_content&view=article&id=336&mode=0&fil=&ox=&cd=09TB&type=&inv=&en=&vn=&ran=0.9122891888036086